CLINICAL TRIAL: NCT04222010
Title: Serratus Plain Block Versus Paravertebral Block Versus Serratus Plain Block and Paravertebral Block for Postoperative Pain Following Thoracoscopic Surgery
Acronym: thoracoscopic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2019_843_0051
Record Dates: First submitted 2019-11-28; First posted 2020-01-09 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Anesthesia, Local; Pain, Postoperative
Keywords: Anesthesia, Local; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- serratus loco-regional anesthesia (Experimental): patient who underwent thoracoscopic surgery will be assigned to serratus plane bloc (Ropivacaine 2 mg/mL, 40 mL) and paravertebral placebo bloc (saline, 20 mL)
  Interventions: Drug: loco-regional anesthesia serratus plane bloc (Ropivacaine 2 mg/mL, 40 mL) and paravertebral placebo bloc (saline, 20 mL)
- paravertebral bloc Loco-regional anesthesia (Experimental): patient who underwent thoracoscopic surgery will be assigned to paravertebral bloc (Ropivacaine 4 mg/mL, 20 mL) and serratus plane placebo bloc (saline, 40 mL)
  Interventions: Drug: Loco-regional anesthesia : paravertebral bloc (Ropivacaine 4 mg/mL, 20 mL) and serratus plane placebo bloc (saline, 40 mL)
- serratus and paravertebral bloc Loco-regional anesthesia (Experimental): patient who underwent thoracoscopic surgery will be assigned to serratus plane bloc (Ropivacaine 1,3 mg/mL, 40 mL) and paravertebral bloc (Ropivacaine 1,3 mg/mL, 20 mL)
  Interventions: Drug: Loco-regional anesthesia : serratus plane bloc (Ropivacaine 1,3 mg/mL, 40 mL) and paravertebral bloc (Ropivacaine 1,3 mg/mL, 20 mL)

INTERVENTIONS:
Drug: loco-regional anesthesia serratus plane bloc (Ropivacaine 2 mg/mL, 40 mL) and paravertebral placebo bloc (saline, 20 mL) — Each patient who underwent thoracoscopic surgery will be assigned to one procedure of Loco-regional anesthesia
  Arms: serratus loco-regional anesthesia
Drug: Loco-regional anesthesia : paravertebral bloc (Ropivacaine 4 mg/mL, 20 mL) and serratus plane placebo bloc (saline, 40 mL) — Each patient who underwent thoracoscopic surgery will be assigned to one procedure of Loco-regional anesthesia.
  Arms: paravertebral bloc Loco-regional anesthesia
Drug: Loco-regional anesthesia : serratus plane bloc (Ropivacaine 1,3 mg/mL, 40 mL) and paravertebral bloc (Ropivacaine 1,3 mg/mL, 20 mL) — Each patient who underwent thoracoscopic surgery will be assigned to one procedure of Loco-regional anesthesia.
  Arms: serratus and paravertebral bloc Loco-regional anesthesia

SUMMARY:
Acute and chronic postoperative pain remains a major concern following thoracoscopic surgery. Firstly because pain constitutes a serious concern for patients after surgery, and secondarily because an ineffective control of pain may lead to postoperative morbidity, especially in lung cancer surgery.

To date, several procedures have been described but the best modality of locoregional analgesia for thoracoscopic surgery has not been assessed yet. The main objective of this study is to evaluate efficiency of several validated approaches for preoperative locoregional analgesia, comparing serratus plain block versus paravertebral block versus serratus plain block and paravertebral block for postoperative pain following thoracoscopic surgery.

To this end, the investigators will conduct an interventional prospective monocentric, double blind, compared and randomized study. Previously to thoracoscopic surgery, patients will be randomized in one of the three following arms: serratus plain block, paravertebral block or serratus plain block and paravertebral block combined.

ELIGIBILITY:
Inclusion Criteria:

* adult patient over18 years old
* without guardianship
* video-assisted thoracoscopic surgery with 3 trocars
* No cons-indications to loco-regional anesthesia (allergy, skin condition)

Exclusion Criteria:

* patient under 18 years old
* patient under guardianship
* pregnant
* rejection of consent
* rejection of loco-regional anesthesia
* chronic pain antecedents under morphine medication
* pain assessment impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Pain Visual analog scale (VAS) score at coughing | Immediately after following thoracoscopic surgery
  Visual analogue scales (VAS) are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain.
  Numerical rating scales are similar to analogue scales except that numbers (e.g., 0 to 5) are entered along the scale.
  With category scales, the patient is asked to circle the word that best describes his or her condition (e.g., for pain intensity: None, Moderate, Severe, Unbearable).

SECONDARY OUTCOMES:
Pain Visual analog scale (VAS) score at coughing | H1 = one hour following thoracoscopic surgery
  Visual analogue scales (VAS) are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain.
  Numerical rating scales are similar to analogue scales except that numbers (e.g., 0 to 5) are entered along the scale.
  With category scales, the patient is asked to circle the word that best describes his or her condition (e.g., for pain intensity: None, Moderate, Severe, Unbearable).
Pain Visual analog scale (VAS) score at coughing | H3 = 3 hours following thoracoscopic surgery
  Visual analogue scales (VAS) are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain.
  Numerical rating scales are similar to analogue scales except that numbers (e.g., 0 to 5) are entered along the scale.
  With category scales, the patient is asked to circle the word that best describes his or her condition (e.g., for pain intensity: None, Moderate, Severe, Unbearable).
Pain Visual analog scale (VAS) score at coughing | H6 = 6 hours following thoracoscopic surgery
  Visual analogue scales (VAS) are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain.
  Numerical rating scales are similar to analogue scales except that numbers (e.g., 0 to 5) are entered along the scale.
  With category scales, the patient is asked to circle the word that best describes his or her condition (e.g., for pain intensity: None, Moderate, Severe, Unbearable).
Pain Visual analog scale (VAS) score at coughing | Day1 = one day following thoracoscopic surgery
  Visual analogue scales (VAS) are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain.
  Numerical rating scales are similar to analogue scales except that numbers (e.g., 0 to 5) are entered along the scale.
  With category scales, the patient is asked to circle the word that best describes his or her condition (e.g., for pain intensity: None, Moderate, Severe, Unbearable).
Pain Visual analog scale (VAS) score at coughing | Day2 = two days following thoracoscopic surgery
  Visual analogue scales (VAS) are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain.
  Numerical rating scales are similar to analogue scales except that numbers (e.g., 0 to 5) are entered along the scale.
  With category scales, the patient is asked to circle the word that best describes his or her condition (e.g., for pain intensity: None, Moderate, Severe, Unbearable).
Pain Visual analog scale (VAS) score at coughing | Day3 = 3 days following thoracoscopic surgery
  Visual analogue scales (VAS) are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain.
  Numerical rating scales are similar to analogue scales except that numbers (e.g., 0 to 5) are entered along the scale.
  With category scales, the patient is asked to circle the word that best describes his or her condition (e.g., for pain intensity: None, Moderate, Severe, Unbearable).

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Berna, Pr, Principal Investigator — CHU Amiens; Emmanuel Lorne, Pr, Principal Investigator — CHU Amiens; Alex Fourdrain, MD, Principal Investigator — CHU Amiens; Florent Leviel, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leviel F, Fourdrain A, Delatre F, De Dominicis F, Lefebvre T, Bar S, Alshatri HY, Lorne E, Georges O, Berna P, Dupont H, Meynier J, Abou-Arab O. S erratus anterior plane block alone, paravertebral block alone and their combination in video-assisted thoracoscopic surgery: the THORACOSOPIC double-blind, randomized trial. Eur J Cardiothorac Surg. 2024 Mar 29;65(4):ezae082. doi: 10.1093/ejcts/ezae082. PMID 38548664